CLINICAL TRIAL: NCT01852305
Title: Would A New Pathway Managing Obstructive Sleep Apnea in Bariatric Surgical Patients Be Safe and Cost-effective?
Brief Title: Obstructive Sleep Apnea in Bariatric Surgical Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to lack resources
Sponsor: University Health Network, Toronto (Other)
Collaborators: Unity Health Toronto (Other); Michael Garron Hospital (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 27/2/2013
Record Dates: First submitted 2013-04-29; First posted 2013-05-13 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Continuous positive airway pressure (CPAP); Oximetry; Bariatric Surgery; Anesthesia; Oxygen desaturation index (ODI)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lab Sleep Study (group 1) (Experimental): The patients in the Sleep Study group will be referred to a sleep medicine specialist who is part of the Bariatric Surgery Psychosocial Program. In the Sleep Study group, patients will undergo sleep studies overnight in a sleep laboratory. At the same time, they will also wear the oximeter wristwatch to measure overnight oximetry.
  Interventions: Other: Lab Sleep Study Group
- Oximetry group (group 2) (Active Comparator): The patients in the Oximetry group will undergo overnight pulse oximetry. The patients with ODI>10 events/hour will be referred to the sleep medicine specialist.A split- night polysomnography(PSG) will be employed to confirm obstructive sleep apnea OSA) diagnosis. The 1st part of the night will be a sleep study and depending on AHI, CPAP titration will be done for the 2nd part of the night.
  Interventions: Device: Oximetry

INTERVENTIONS:
Other: Lab Sleep Study Group — Patients in this group will under go lab sleep study overnight at the sleep clinic.If the patient has severe sleep apnea (AHI>30) or moderate sleep apnea (AHI>15 to <30) with significant co-morbidities (e.g. cardiovascular disease, diabetes), CPAP treatment will be recommended. For mild sleep apnea (AHI>5 to <15) or moderate sleep apnea without significant co-morbidities, CPAP will not be required. If patient is not able to tolerate or refuses CPAP, dental device and positional therapy will be recommended.
  Other Names: Lab polysomnography study
  Arms: Lab Sleep Study (group 1)
Device: Oximetry — The patients in the Oximetry group will undergo overnight pulse oximetry. The patients with ODI>10 events/hour will be referred to the sleep medicine specialist.A split- night PSG will be employed to confirm OSA diagnosis. The 1st part of the night will be a sleep study and depending on AHI, CPAP titration will be done for the 2nd part of the night
  Other Names: oximeter/group 2
  Arms: Oximetry group (group 2)

SUMMARY:
Purpose:

The purpose of this study is to develop a novel pathway to decrease the cost and waiting time to manage bariatric surgical patients with obstructive sleep apnea.

Hypotheses:

Compared to the current perioperative pathway, the proposed novel pathway incorporating overnight oximetry and perioperative sleep apnea precautions is safe and more cost effective for evaluating and managing obstructive sleep apnea in the bariatric surgical patients.

To decrease the cost and waiting time, we proposed a novel perioperative pathway to manage obstructive sleep apnea in the bariatric patients. In this pathway, the patient will be screened by the STOP-Bang questionnaire. The recruited patients will be randomized into two groups:

The STOP-Bang questionnaire score is ≥4 then you will be assigned to any one of these groups

* sleep study group (group 1) or
* oximetry group (group 2).

DETAILED DESCRIPTION:
The potential patients will be screened by the STOP-Bang questionnaire. Those with a score ≥4 will be randomized into Sleep Study group or Oximetry group. The patients in the Sleep Study group will be referred to a sleep medicine specialist who is part of the Bariatric Surgery Psychosocial Program. In the Sleep Study group, patients will undergo sleep studies overnight in a sleep laboratory. At the same time, they will also wear the oximeter wristwatch to measure overnight oximetry. Depending on the sleep study results and medical history, a decision will be made regarding therapeutic options. If the patient has severe sleep apnea (AHI>30) or moderate sleep apnea (AHI>15 to <30) with significant co-morbidities (e.g. cardiovascular disease, diabetes), CPAP treatment will be recommended. For mild sleep apnea (AHI>5 to <15) or moderate sleep apnea without significant co-morbidities, CPAP will not be required. If patient is not able to tolerate or refuses CPAP, dental device and positional therapy will be recommended.

The patients in the Oximetry group will undergo overnight pulse oximetry. The patients with ODI>10 events/hour will be referred to the sleep medicine specialist. Since the patients with ODI>10 had a high probability 69%) to have moderate and severe OSA. A split- night PSG will be employed to confirm OSA diagnosis and to titrate CPAP with in patients with ODI>10. The 1st part of the night will be a sleep study and depending on AHI, CPAP titration will be done for the 2nd part of the night. Compared to Sleep Study group, only one night instead of two nights of sleep studies is needed in patients with ODI>10 events/hour. The patients with ODI ≤ 10 events/h will undergo surgery with routine care plus sleep apnea perioperative precautions.

ELIGIBILITY:
Inclusion/Exclusion criteria: The patients who meet the following criteria will be recruited.

* Patients undergoing bariatric surgery with American Society of Anaesthesiologists (ASA) score 1-4 will be approached.
* The patients with any of the following conditions will be excluded:

  1. Unable or not willing to give an informed consent;
  2. Potential problems with EEG;
  3. Patients with diagnosed OSA.
  4. Patients having sleep study before.
  5. Age: < 18 years having sleep study before. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2013-04; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
The average cost for obstructive sleep apnea management | 30 days after surgery
  The average cost for obstructive sleep apnea management during the period from the initial assessment visit to 30 days after surgery.
The incidence of postoperative adverse events | 30 days after surfery
  The composite incidence of postoperative adverse events

SECONDARY OUTCOMES:
Number of visits to the health care professionals | 1 year
  The secondary outcomes will be the number of visits to MDs, emergency and the length of hospital stay within the same period.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS FRCPC, Principal Investigator — University Health Network,University of Toronto; David Mazer, MD, Principal Investigator — St. Michael's Hospital, University of Toronto; James Kulchyk, MD, Principal Investigator — Toronto East General Hospital, University of Toronto
Locations (1):
- 399 Bathurst St.,Toronto Western Hopsital, Preadmission Clinic, Dept. of Anesthesia, Toronto, Ontario, Canada